CLINICAL TRIAL: NCT05115331
Title: 1-2 PUNCH: Palliative UNConventional Hypofractionation Trial for Metastatic Bone Disease
Brief Title: Palliative UNConventional Hypofractionation Trial for Metastatic Bone Disease
Acronym: 1-2 PUNCH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Timothy Struve, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCC-RT-21-01
Record Dates: First submitted 2021-10-15; First posted 2021-11-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Bone Tumor
Keywords: Metastatic Bone Disease
MeSH Terms: conditions — Bone Neoplasms; Bone Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Radiation Dose (Active Comparator): 8 Gy in a single fraction
  Interventions: Radiation: Conventional Radiation Dose
- Experimental Radiation Dose (Experimental): 16 Gy in 2 fractions
  Interventions: Radiation: Experimental Radiation Dose

INTERVENTIONS:
Radiation: Experimental Radiation Dose — 16 Gy in 2 fractions
  Arms: Experimental Radiation Dose
Radiation: Conventional Radiation Dose — 8 Gy in a single fraction
  Arms: Conventional Radiation Dose

SUMMARY:
This is a randomized Phase III study evaluating the efficacy of hypofractionated and dose-escalated palliative radiation therapy in metastatic bone disease (MBD). Patients will be randomized 1:1 to the conventional (8 Gy in a single fraction) and experimental (16 Gy in 2 fractions) groups with baseline and subsequent assessment of both pain and quality of life metrics.

DETAILED DESCRIPTION:
Metastatic Bone Disease (MBD) has been demonstrated to be a common clinical problem, and often presents with severe, if not debilitating pain. This often proceeds to affect a patient's emotional and even global functioning. Radiation therapy is an effective treatment commonly used in the palliation of these metastatic lesions, and improvements in QOL scores are associated with response to radiotherapy treatment. Although both 30 Gy/10 fractions and 8 Gy in a single fraction are considered standard of care in the palliative setting, single fraction treatment is associated with increased rates of local failure and retreatment. Considering that patients with MBD often have life-limiting disease, and frequently have great difficulty with undergoing extended radiotherapy treatments, there is a significant unmet need for palliative treatments that are effective, safe, timely, and provide a durable local tumor and pain control. The investigators hypothesize that utilizing a fractionation scheme with an escalated biologically equivalent dose will result in a higher proportion of patients responding to treatment, and will also lead to more durable responses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed history of solid cancer malignancy (including small cell lung cancer).
2. Patients must have 1-3 new or newly painful metastatic lesions to bone as defined by CT scan, MRI, or PET scan. Lesions must be located in a long bone, pelvis/hip, spine, sacrum, or ribs. A lesion is "new" if it has occurred since any previous imaging, or if new cancer diagnosis, or new at presentation. A newly painful lesion is one that had been visible on previous imaging, but was either asymptomatic or minimally painful so that no treatment was pursued.
3. There must be clearly attributable pain associated with the 1-3 new metastatic bone lesion(s) as documented on the Brief Pain Inventory and per investigator's determination that these imaging findings are consistent with the patient's described BPI pain from metastatic lesion(s).
4. Age ≥18 years.
5. ECOG performance status ≤3 or (Karnofsky ≥40%, see Appendix A).
6. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial in the opinion of the investigator.
7. Ability to understand and the willingness to sign written informed consent.

Exclusion Criteria:

1. Patients who have had or will have chemotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to commencing study RT. Patients undergoing treatment with hormonal or endocrine therapies will be eligible for this trial and may continue these through study radiotherapy.
2. Patients with widespread metastatic disease, such that in the opinion of the PI would preclude an investigator from determining the origin of bone disease-related pain and/or response to palliative treatment.
3. Patients who are receiving any other investigational agents. Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI.
4. Patients with complicated bone metastases, defined as having at least one or more of the following criteria:

   1. Nerve root compression
   2. Prior radiation to the spinal cord at that bone level
   3. Impending (score of 9 or more on Mirel's Criteria) or existing pathologic fracture
   4. Spinal cord compression
   5. cauda equina syndrome
5. Patients who have been previously radiated to the primary anatomic site for which they are being considered for this trial, or have had surgical fixation of the site. However, patients may have undergone previous courses of radiotherapy to a primary site or separate site of metastatic disease if in the opinion of the investigator the patient will be able to tolerate palliative RT.
6. Patients with uncontrolled intercurrent illness.
7. Pregnant women are excluded from this study.
8. Life expectancy of under 3 months in the opinion of the treating investigator.
9. Liquid malignancies, including myeloma, lymphoma.
10. Judgment by the investigator that the patient is unsuitable to participate in the study or the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Pain Response measured by the Brief Pain Inventory | 1 month post radiation completion.
  A primary objective evaluate the efficacy of the addition of a second 8 Gy fraction administered 1 week following the standard 8 Gy treatment currently utilized for palliation of symptomatic bone metastases in solid cancers, as measured by pain response at 1 month. The primary endpoint for this objective is pain response which will be determined using the Brief Pain Inventory (BPI) at one month.
Pain Response measured by the Bone Mets Pain scale | 1 month post radiation completion.
  A primary objective evaluate the efficacy of the addition of a second 8 Gy fraction administered 1 week following the standard 8 Gy treatment currently utilized for palliation of symptomatic bone metastases in solid cancers, as measured by pain response at 1 month. The primary endpoint for this objective is pain response which will be classified using the International Consensus on Palliative Radiation for Future Trials on Bone Mets, which is a 4-point scale ranging from complete response to pain progression. Pain relief as measured by this scale and daily oral morphine equivalents (OME) will be graded at 1 month.
Safety through 30 days post-radiation | 30 days post radiation completion.
  A second primary objective is to characterize the safety profile and adverse events (AE) of dose-escalated palliative radiotherapy. The primary endpoint for this objective is Adverse events will be described and coded based upon the NCI CTCAE v5.0 through 30 days after end of a subject's treatment.

SECONDARY OUTCOMES:
Time to pain relief | 2, 3, and 6 months after completion of radiation treatment.
  A secondary objective is to determine time to maximal pain relief, and to determine pain response at 2, 3, and 6 months. Pain response at 2, 3, and 6 months will be assessed using the Brief Pain Inventory (BPI), and classified using the International Consensus on Palliative Radiation for Future Trials on Bone Mets; as well as daily oral morphine equivalents (OME). Time to maximal pain relief will be determined from BPI questionnaires and International Consensus on Palliative Radiation for Future Trials on Bone Mets scale data.
Quality of Life (EORTC QLQ-C30) at Baseline, 1, 3, and 6 months post treatment | Baseline, 1, 3, and 6 months post radiation treatment.
  Another secondary objective is to evaluate the impact of standard and dose-escalated arms of palliative radiotherapy on quality of life. Quality of life data will be obtained via European Organisation for Research and Treatment of Cancer Quality of Life Cancer Patients (EORTC QLQ-C30 (version 3)) at baseline and 1-, 3-, and 6-months post-treatment.
Quality of Life (EORTC QLQBM22) at Baseline, 1, 3, and 6 months post treatment | Baseline, 1, 3, and 6 months post radiation treatment.
  Another secondary objective is to evaluate the impact of standard and dose-escalated arms of palliative radiotherapy on quality of life. Quality of life data will be obtained via European Organisation for Research and Treatment of Cancer Quality of Life Bone Metastases (EORTC QLQBM22) at baseline and 1-, 3-, and 6-months post-treatment.
Overall survival through 2 years post-treatment. | 2 years post treatment.
  Another secondary objective is to determine differences in overall survival between subjects receiving standard and dose-escalated palliative radiotherapy. Overall survival (OS) data from the date of completion of radiation therapy will be obtained from departmental records and electronic medical records through 2 years post end of radiation treatment.
Retreatment rates through 2 years post-treatment. | 2 years post treatment.
  Another secondary objective is to determine differences in retreatment rates between subjects receiving standard and dose-escalated palliative radiotherapy. Retreatment rates data from the date of completion of radiation therapy will be obtained from departmental records and electronic medical records through 2 years post end of radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Struve, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No